CLINICAL TRIAL: NCT03320148
Title: Determining the Impact of a New Physiotherapist Led Primary Care Model for Back Pain: A Pilot Cluster Randomized Controlled Trial
Brief Title: Determining the Impact of a New Physiotherapist Led Primary Care Model for Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Jordan Miller, PT, PhD, Assistant Professor, School of Rehabilitation Therapy, Queen's University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 6021536
Record Dates: First submitted 2017-10-16; First posted 2017-10-25 (Actual); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: Back Pain
MeSH Terms: conditions — Back Pain

STUDY DESIGN:
Intervention Model Description: This is a pilot cluster randomized controlled trial randomizing 4 sites to the PT-led primary care model for back pain or usual care model
Masking Description: Due to the nature of the new model of care and comparison, it is not possible to blind the patients or health care providers. Since the primary outcomes are self-reported outcome measures, the assessor is also not blind to the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physiotherapist-led primary care model for back pain (Experimental): The PT-led primary care model for back pain will involve incorporating a PT within the primary care team at the first point of contact for people with back pain at no cost to the patient. Patients in this model will be given the choice of seeing the PT or family doctor. They will be encouraged to book with the PT except when the primary reason for visit is for medication renewals or when the patient has additional health concerns that need attention from their physician in the same visit. There will be 4 key components of the PT led primary care intervention: 1) Initial assessment and screening; 2) Brief individualized intervention at the first visit; 3) Health services navigation; 4) Providing additional PT care for people with an unmet need.
  Interventions: Behavioral: Physiotherapist-led primary care model for back pain
- Usual care (Active Comparator): The physician led primary care intervention will be unstandardized to best reflect standard clinical practice in Canada. This usually includes a visit to a primary care physician, who would perform a history and physical examination, provide LBP education, and prescribe medications and/or refer based on their assessment findings and patient preferences.
  Interventions: Other: Usual care

INTERVENTIONS:
Behavioral: Physiotherapist-led primary care model for back pain — 1. Assessment and screening: taking a history; screening for red flags, comorbidities, and risk factors of ongoing pain and disability; physical examination
  2. Brief individualized intervention at the first visit: effective communication, cognitive reassurance, a few exercises, and advice/strategies to stay active.
  3. Health services navigation: PT assistance with navigating healthcare services based on the assessment findings. First, red-flags requiring emergency or urgent referrals. Next, comorbid conditions that would benefit from care from other healthcare providers. Finally, referral to PT (if appropriate).
  4. Providing additional physiotherapy care to people with an unmet need: Additional physiotherapy care will be provided to patients who have an identified need for physiotherapy but no physiotherapy coverage through private or government health insurance plans.
  Arms: Physiotherapist-led primary care model for back pain
Other: Usual care — The physician led primary care intervention will be unstandardized to best reflect standard clinical practice in Canada.
  Arms: Usual care

SUMMARY:
This is a pilot cluster randomized controlled trial to determine the feasibility of a cluster randomized trial to evaluate the individual and health system impact of implementing a new physiotherapist-led primary care model for back pain in Canada.

DETAILED DESCRIPTION:
This study aims to determine the feasibility of conducting a cluster randomized trial in primary care settings in Ontario to evaluate the individual health outcomes and health system impact of implementing a new physiotherapist-led primary care model for people with back pain. The primary purpose of this pilot study is to determine the feasibility including recruitment and retention of primary care teams (sites) and patient participants, carrying out the assessment procedures, and implementing the physiotherapist-led primary care intervention including training the physiotherapist to adopt this role.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 years and over) with back pain of any duration
* Seeking primary care for back pain at a participating site
* Primary care visit may be a first or repeat visit

Exclusion Criteria:

* Patients who do not consent to participation
* Patients who report being unable to understand, read, and write English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-09-20 (Actual); Primary Completion 2019-01-15 (Actual); Study Completion 2019-01-15 (Actual)

PRIMARY OUTCOMES:
Recruitment of primary care teams | Baseline
  Ability to recruit four primary care teams (Family Health Teams or Community Health Centres) to paricipate
Recruitment of patient participants | Baseline to 14 weeks
  Recruitment rate (participants/week) or total number of participants recruited in 14 weeks
Assessment completion | Baseline, 6-week 12-week, 6,9,12 month follow-up. The primary time point for this assessment is 12-week follow-up.
  Percentage of all assessment items completed by participants completing each assessment
Retention of patient participants | Retention of participants at 6-week, 12-week, 6, 9, and 12-month follow-up assessments. The primary timeline for this outcome is 12-month follow-up.
  Attrition rate
Physiotherapist confidence in carrying out the interventions | Baseline
  The PT will rate his/her confidence in each component of the intervention after the training on a scale from 0-10 with higher scores indicating greater confidence in carrying out that component of the intervention.
Treatment fidelity | 6-week follow-up
  Treatment fidelity will be measured by consistency with the intervention described in the protocol measured through an intervention checklist completed by the physiotherapist and an audit of the EMR notes.

SECONDARY OUTCOMES:
Self-reported disability | Baseline, 6-week, 12-week, 6-month, 9-month, and 12-month follow-up
  measured using the Roland Morris Disability Questionnaire (0 to 24 with higher scores indicating greater disability)
Self-reported pain intensity | Baseline, 6-week, 12-week, 6-month, 9-month, and 12-month follow-up
  measured using a numeric pain rating scale from 0 to 10 with higher scores indicating greater pain intensity (measured at rest, during walking, and during a lifting task)
Health Related Quality of Life | Baseline, 6-week, 12-week, 6-month, 9-month, and 12-month follow-up
  measured using the EuroQoL-5D-5L (0 to 100 with greater scores indicating greater self-reported health related quality of life)
Global rating of change | Baseline, 6-week, 12-week, 6-month, 9-month, and 12-month follow-up
  measured using an 11-point scale (-5 to +5 with negative scores indicating a worsening of physical functioning related to back pain and positive scores indicating an improvement of physical functioning related to back pain)
Satisfaction with health care | Baseline, 6-week, 12-week, 6-month, 9-month, and 12-month follow-up
  measured using an 11-point scale(-5 to +5 with negative scores indicating a dissatisfaction with health care received and positive scores indicating satisfaction with health care received)
Catastrophic Thinking | Baseline, 6-week, 12-week, 6-month, 9-month, and 12-month follow-up
  measured using the Pain Catastrophizing Scale (0 to 52 with higher scores indicating greater catastrophic thinking)
Depressive symptoms | Baseline, 6-week, 12-week, 6-month, 9-month, and 12-month follow-up
  measured using the 9-item Patient Health Questionnaire (PHQ-9) (0 to 27 with greater scores indicating increased depressive symptoms)
Adverse events | Baseline, 6-week, 12-week, 6-month, 9-month, and 12-month follow-up
  measured using an adverse events questionnaire that asks 1) if the patient has experienced any adverse events as a result of the treatments received (yes/no); 2) how long the event lasted (hours or days); 3) how severe the adverse event was (0-10 scale); 4) what adverse events were experienced.
Health care accessibility | Baseline, 6-week, 12-week, 6-month, 9-month, and 12-month follow-up
  Percentage of patients receiving care within 48 hours.
Health care accessibility | Baseline, 6-week, 12-week, 6-month, 9-month, and 12-month follow-up
  Percentage of patients who score medium or high risk on the STarT Back tool who receive physiotherapy care.
Health care utilization | Baseline, 6-week, 12-week, 6-month, 9-month, and 12-month follow-up
  All health care visits (aggregated and dis-aggregated) including: primary care visits, emergency department visits, hospitalizations, surgeries, consultations with other health care providers, diagnostic imaging, medications, and other care received by the patient
Costs (piloted for a cost utility analysis in a future trial) | Baseline, 6-week, 12-week, 6-month, 9-month, and 12-month follow-up
  Includes all health care costs plus societal costs using a human capital approach for loss of productivity
Medications prescribed | Baseline, 6-week, 12-week, 6-month, 9-month, and 12-month follow-up
  Measured as a process outcome
Diagnostic imaging ordered | Baseline, 6-week, 12-week, 6-month, 9-month, and 12-month follow-up
  Measured as a process outcome
referrals to other health care providers made | Baseline, 6-week, 12-week, 6-month, 9-month, and 12-month follow-up
  Measured as a process outcome
notes made by primary care provider to employers or insurers | Baseline, 6-week, 12-week, 6-month, 9-month, and 12-month follow-up
  Measured as a process outcome

CONTACTS AND LOCATIONS:
Overall Officials: Jordan Miller, PhD, Principal Investigator — Queen's University
Locations (1):
- Queen's University, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data from this pilot study. This data will be used to inform the protocol for a fully powered cluster randomized trial.

REFERENCES:
- [Derived] Miller J, Barber D, Donnelly C, French S, Green M, Hill J, MacDermid J, Marsh J, Norman K, Richardson J, Taljaard M, Wideman T, Cooper L, McPhee C. Determining the impact of a new physiotherapist-led primary care model for back pain: protocol for a pilot cluster randomized controlled trial. Trials. 2017 Nov 9;18(1):526. doi: 10.1186/s13063-017-2279-7. PMID 29121989